CLINICAL TRIAL: NCT05463497
Title: A Randomized, Open-label, Multiple-dose, 2x3 Crossover Clinical Trial to Investigate the Pharmacokinetic Drug Interaction of JW0201 and C2103 or C2104 After Oral Administration in Healthy Adults
Brief Title: To Evaluate the Pharmacokinetic Drug Interactions, Safety and Drug Tolerance in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: JW21101
Record Dates: First submitted 2022-07-03; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: A randomized, open-label, multiple-dose, 2x3 crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1(N=10) (Other): Treatment A for Period 1 Treatment C for Period 2 Treatment B for Period 3
  *Washout period : No washout period between period 1 and 2, more than 7 days between period 2 and 3
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Group 2(N=10) (Other): Treatment B for Period 1 Treatment A for Period 2 Treatment C for Period 3
  *Washout period : more than 7 days between period 1 and 2, no washout period between period 2 and 3
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Group 3(N=10) (Other): Treatment A for Period I Treatment E Treatment D
  *Washout period : No washout period between period 1 and 2, more than 7 days between period 2 and 3
  Interventions: Drug: Treatment A; Drug: Treatment D; Drug: Treatment E
- Group 4(N=10) (Other): Treatment D for Period 1 Treatment A for Period 2 Treatment E for Period 3
  *Washout period : more than 7 days between period 1 and 2, no washout period between period 2 and 3
  Interventions: Drug: Treatment A; Drug: Treatment D; Drug: Treatment E

INTERVENTIONS:
Drug: Treatment A — JW0201: single administration, Tablet, Oral, BID for 5 days
Drug: Treatment B — C2103: single administration, Tablet, Oral, BID for 5 days
  Arms: Group 1(N=10); Group 2(N=10)
Drug: Treatment C — JW0201 and C2103 : combination administration, Tablet, Oral, BID for 5 days
  Arms: Group 1(N=10); Group 2(N=10)
Drug: Treatment D — C2104 : single administration, Tablet, Oral, QD for 5 days
  Arms: Group 3(N=10); Group 4(N=10)
Drug: Treatment E — JW0201 and C2104 : combination administration, JW0201 twice a day and C2104 once a day for 5days
  Arms: Group 3(N=10); Group 4(N=10)

SUMMARY:
A randomized, open-label, multiple-dose, 2x3 crossover clinical trial to investigate the pharmacokinetic drug interaction of JW0201 and C2103 or C2104 after oral administration in healthy adults

DETAILED DESCRIPTION:
1. To evaluate the pharmacokinetic characteristics, safety, and drug tolerance of combined administration JW0201 and C2103 compared to the case of each single administration in healthy adults.
2. To evaluate the pharmacokinetic characteristics, safety, and drug tolerance of combined administration JW0201 and C2104 compared to the case of each single administration in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Subjects does not meet the Inclusion Criteria

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | up to 12hour(or 24hour) after administration
  Cmax,ss of each drug
AUCτ,ss | up to 12hour(or 24hour) after administration
  AUCτ,ss of each drug

SECONDARY OUTCOMES:
Cmin,ss | up to 12hour(or 24hour) after administration
  Cmin,ss of each drug
Tmax,ss | up to 12hour(or 24hour) after administration
  Tmax,ss of each drug
CLss/F | up to 12hour(or 24hour) after administration
  CLss/F of each drug
Vdss/F | up to 12hour(or 24hour) after administration
  Vdss/F of each drug
fluctuation | up to 12hour(or 24hour) after administration
  fluctuation of each drug

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, PI, Principal Investigator — Jeonbuk National University Hospita
Locations (1):
- Jeonbuk National University Hospita, Jeonju, Jeollabuk-do, South Korea